CLINICAL TRIAL: NCT04927884
Title: Open-Label Phase 1b/2 Study of Sacituzumab Govitecan-Hziy Plus Chemoimmunotherapy for the Treatment of Subjects With Advanced Triple-Negative Breast Cancer After Prior Therapy
Brief Title: A Study of Sacituzumab With Chemoimmunotherapy to Treat Advanced Triple-Negative Breast Cancer After Prior Therapies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.058
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Advanced Triple Negative Breast Cancer
Keywords: Chemoimmunotherapy; Stage IV TNBC; Sacituzumab; N-803; PD-L1 t-haNK; Cyclophosphamide
MeSH Terms: interventions — ALT-803; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Sacituzumab plus chemoimmunotherapy (cyclophosphamide, N-803, and PD-L1 t-haNK)
  Interventions: Biological: N-803; Biological: PD-L1 t-haNK; Drug: Sacituzumab Govitecan-Hziy; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: N-803 — Dose: 15 μg/kg subcutaneously (SC)
  Frequency: administered on Day 8 of each cycle (every 3 weeks)
Biological: PD-L1 t-haNK — Dose: ~2 × 10^9 cells intravenously (IV)
  Frequency: administered on Days 1 and 8 of each cycle (every 3 weeks)
Drug: Sacituzumab Govitecan-Hziy — Phase 1b:
  Dose level 1: Sacituzumab govitecan-hziy (7.5 mg/kg IV) Dose level 2: Sacituzumab govitecan-hziy (10 mg/kg IV) Dose level -1 (if needed): Sacituzumab govitecan-hziy (5.0 mg/kg IV)
  Phase 2: Dose based on Phase 1b Recommended Phase 2 Dose (IV)
  Frequency: administered on Days 1 and 8 of each cycle (every 3 weeks)
Drug: Cyclophosphamide — Dose: 25 mg capsules taken twice per day by mouth (PO)
  Frequency: to be taken Days 1-15 and 15-19 of each cycle (every 3 weeks)

SUMMARY:
This is a phase 1b/2 open-label study to evaluate the safety and efficacy of sacituzumab govitecan-hziy in combination with chemoimmunotherapy (cyclophosphamide, N-803, and PD-L1 t-haNK) in subjects with Triple Negative Breast Cancer (TNBC) after at least 2 prior treatments for metastatic disease.

DETAILED DESCRIPTION:
In part 1 of phase 1b, 3 to 6 subjects will be sequentially enrolled starting at dose level 1 and will be assessed for dose limiting toxicities (DLTs). Dose level cohorts for sacituzumab govitecan-hziy are as follows:

* Dose level 1: Sacituzumab govitecan-hziy (7.5 mg/kg IV)
* Dose level 2: Sacituzumab govitecan-hziy (10 mg/kg IV)
* Dose level 1 (if needed): Sacituzumab govitecan-hziy (5.0 mg/kg IV)

In part 2 of phase 1b, dose expansion will occur when the RP2D has been determined. An additional 4 subjects may be enrolled, for a total of up to 10 subjects at the RP2D. Following part 2 of the phase 1b portion of the study, the Safety Review Committee (SRC) will meet to determine if enrollment into phase 2 should proceed.

In the phase 2 portion of the study, 22 subjects will be enrolled at the RP2D in the first stage of Simon's two stage optimal design. If ≥ 9 of 22 subjects exhibit a confirmed response, the study will proceed to the second stage.

If the study proceeds to the second stage, an additional 41 subjects will be enrolled for a total of 63 subjects in the phase 2. If ≥ 27 of the 63 subjects exhibit a confirmed response, the combination therapy will be considered for further development.

All subjects may receive up to 17 cycles (ie, 51 weeks) of treatment administered in 3-week cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically confirmed stage IV TNBC. Subjects must have had at least 2 prior treatments for TNBC. TNBC is defined as breast cancer that lacks estrogen receptor (ER) and progesterone receptor (PgR) expression (both ≤ 1% of tumor cell nuclei), and human epidermal growth factor receptor 2 (HER2) overexpression and/or amplification (IHC 0 or 1+, or IHC 2+ and fluorescence in situ hybridization [FISH]-), according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guideline criteria, as evaluated by local institutions.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm and/or non-measurable disease evaluable in accordance with RECIST V1.1.
6. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
7. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception while on study and for at least 5 months after the last dose of study treatment. Non-sterile male subjects must agree to use a condom while on study and for up to 5 months after the last dose of study treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), oral contraceptives, and abstinence.

Exclusion Criteria:

1. Have previously received or are currently receiving treatment with sacituzumab govitecan-hziy.
2. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
3. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
4. History of organ transplant requiring immunosuppression.
5. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
6. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) < 1500 cells/mm3.
   2. Platelet count < 75,000 cells/mm3.
   3. Hemoglobin < 9 g/dL.
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase (ALP) levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
7. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
8. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
9. Known hypersensitivity to any component of the study medication(s).
10. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
11. Known uridine diphosphate-glucuronosyl transferase 1A1 (UGT1A1) gene polymorphism resulting in reduced function.
12. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
13. Concurrent participation in any interventional clinical trial.
14. Pregnant and nursing women. A negative serum pregnancy test during screening and a negative pregnancy test within 72 hours prior to the first dose must be documented before study drug is administered to a female subject of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Reddy, MD, Study Director — ImmunityBio, Inc.
Locations (1):
- Hoag Memorial Hospital, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
Groups:
- Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects: Sacituzumab plus chemoimmunotherapy (cyclophosphamide, N-803, and PD-L1 t-haNK) Sacituzumab govitecan-hziy 7.5 mg/kg IV for all subjects N-803: Dose: 15 μg/kg subcutaneously (SC)
  Frequency: administered on Day 8 of each cycle (every 3 weeks)
  PD-L1 t-haNK: Dose: ~2 × 10^9 cells intravenously (IV)
  Frequency: administered on Days 1 and 8 of each cycle (every 3 weeks)
Period: Overall Study
Arm/Group | Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects
Started | 3
Completed | 1
Not Completed | 2
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Histologically confirmed stage IV TNBC. Subjects must have had at least 2 prior treatments for TNBC [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Time Frame: 30 days after last dose, up to 65 weeks and 5 days
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Number of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 30 days after last dose, up to 65 weeks and 5 days weeks or until resolution or stabilization for nonserious grade 3 or 4 AEs and SAEs, whichever is longer.
Description: Only the Phase 1b portion of the study enrolled participants at the 7.5 mg/kg Sacituzumab Govitecan-Hziy dose level. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
Arm/Group | Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects (N=3)
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Central nervous system lesion (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan-hziy 7.5 mg/kg IV for All Subjects (N=3)
Nausea (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Injection site pain (General disorders) | 2
Injection site pruritus (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Feeling jittery (General disorders) | 1
Gait disturbance (General disorders) | 1
Injection site erythema (General disorders) | 1
Peripheral swelling (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Dyspnoea (Metabolism and nutrition disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Central nervous system lesion (Nervous system disorders) | 1
Cognitive linguistic deficit (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Lymphoedema (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment. Only the safety data is provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04927884/Prot_SAP_000.pdf